CLINICAL TRIAL: NCT03079973
Title: A Randomized, Doubleblind, Vehicle-controlled, Parallel-group Trial to Assess the Efficacy, Safety and Tolerability of P-3073 for Topical Treatment of Nail Psoriasis
Brief Title: Study to Evaluate the Efficacy and Safety of P-3073 Nail Solution in the Treatment of Mild to Moderate Psoriatic Fingernail/s
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Project development priorities changed.
Sponsor: Polichem S.A. (Industry)
Collaborators: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PM1440; NCT03209388 (obsolete NCT alias)
Record Dates: First submitted 2017-03-09; First posted 2017-03-15 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Nail Psoriasis
Keywords: Calcipotriene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- P-3073 (Experimental)
  Interventions: Drug: P-3073 (calcipotriene 0.005%)
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle of P-3073

INTERVENTIONS:
Drug: P-3073 (calcipotriene 0.005%) — Topical solution P-3073 (calcipotriene 0.005%) once daily for 24 weeks.
  Arms: P-3073
Drug: Vehicle of P-3073 — Once daily for 24 weeks.
  Arms: Vehicle

SUMMARY:
The objective of this phase III study is to evaluate the efficacy, systemic safety and local tolerability of P-3073 (calcipotriene 0.005%) nail solution in patients with mild to moderate psoriatic fingernail/s.

DETAILED DESCRIPTION:
This phase III study versus vehicle will be conducted to confirm the clinical efficacy and safety of P-3073 in patients affected by isolated psoriatic nail(s) and/or those with psoriatic nails and concomitant mild-to-moderate plaque psoriasis.

The evaluation of the primary endpoint will be made using the Nail Psoriasis Severity Index (NAPSI).

The secondary objectives will be:

* To assess if the topical treatment with P-3073 is able to improve the quality of life and discomfort in patients with psoriatic fingernail.
* To assess the safety and tolerability of topical P-3073 in the treatment of psoriatic fingernail.

The study consists of two arms comparing P-3073 (calcipotriene 0.005%) and vehicle. Eligible patients will be randomized to either P-3073 or placebo in a 1:1 ratio, stratified by their target nail NAPSI severity at screening.

The study population will include at least 470 patients (235 for each group) with nail psoriasis (fingernails) of the matrix and/or of the nail bed in at least one fingernail.

The total duration of the trial for each patient will be approximately 29 weeks (from Screening to Follow-up). During the 24 weeks of the treatment period, patients will apply the assigned treatment to all affected psoriatic fingernails once daily.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent before starting any study related procedure.
* Patients ages ≥ 18 and ≤ 80 years old.
* Men or women.
* Outpatients.
* Patients with mild to moderate psoriatic fingernail/s, defined as fingernail/s with matrix psoriasis NAPSI score and/or bed psoriasis NAPSI score ≥ 1 and ≤ 3 at baseline. The sum of the scores for each nail should range between 1 and 6.
* In case of skin involvement, patients with established clinical diagnosis of mild to moderate psoriasis (BSA involvement ≤ 8% or Psoriasis Area Severity Index (PASI) ≤ 10).

Exclusion Criteria:

* Use of any systemic treatment for psoriasis and/or nail psoriasis during the last six months before the screening visit.
* Use of any topical treatment for nail psoriasis on fingernails during the last six months before the screening visit.
* Use of photochemotherapy (phototherapy is allowed) or other forms of radiotherapy during the last four weeks before the screening visit.
* Positive mycology findings (KOH evaluation or culture) obtained in the three months before the screening visit or positive KOH evaluated at the screening visit.
* Patients using nail polish or other nail cosmetic products during last 72 hours prior to study drug application.
* Systemic use of the following therapies for any reason during last three months before the screening visit: immunosuppressives, chemotherapy and corticosteroids (topical use for plaque psoriasis is allowed).
* Consumption of oral Vitamin D or its analogues for any reason during the last three months before the screening visit (Calcipotriene topical use for plaque psoriasis is allowed).
* Patients with a clinically significant history of cardiovascular, renal, neurologic, liver, immunologic or endocrine dysfunction. A clinically significant disease is defined as one that in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease that may influence the results of the study or the patient's ability to participate in the study.
* Patients with a recent history (< 1 year) of myocardial infarction and/or (< 3 years) of heart failure or patients with any cardiac arrhythmia requiring drug therapy.
* History of hypercalcaemia or hypercalciuria.
* History of previous or current malignancy in particular lymphoma, melanoma and/or basal cell carcinoma.
* History of allergic reactions to Calcipotriene or P-3073 excipients.
* Patients unable to understand the procedures and purposes of the study.
* Patients unable or unwilling to accept and meet study requirements.
* Use of an investigational drug or participation in an investigational study within 30 days, or 6 half lives whichever is longer, prior to application of study medication.
* Alcohol or substance abuse.
* AIDS symptoms or any other immunodeficiency.

Additional exclusion criteria for females only:

* Breast-feeding patients.
* Positive urine pregnancy test at screening (performed for all females of child bearing potential or for those in non-surgical post-menopause for less than 1 year).
* Female of childbearing potential having unprotected sexual intercourse with any non-sterile male partner (i.e., a male who has not been sterilized by vasectomy at least 6 months prior to drug application) within 14 days prior to study drug application. Acceptable methods of contraception are the following: condom, diaphragm, intrauterine contraceptive device (placed at least 4 weeks prior to study drug application), pill + condom.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-15 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with clear target nail at Week 24 | Week 24
  Defined as Nail Psoriasis Severity Index (NAPSI) =0

SECONDARY OUTCOMES:
Proportion of affected nails at baseline with NAPSI=0 at Week 24 | Baseline - Week 24
  Defined as affected nails with NAPSI=0
Proportion of patients with clear target nail bed at Week 24 | Baseline - Week 24
  Defined as nail bed in NAPSI=0
Proportion of patients with clear target nail matrix at Week 24 | Baseline - Week 24
  Defined as nail matrix in NAPSI=0

OTHER OUTCOMES:
Proportion of patients with target nail reaching NAPSI-75% | Baseline - Week 24
  Defined as a reduction of ≥75% from baseline NAPSI score
Proportion of affected nails at baseline reaching NAPSI-75% | Baseline - Week 24
  Defined as a reduction of ≥75% from baseline NAPSI score
Change from Baseline in Total NAPSI at Week 24 | Baseline - Week 24
  Defined as change in Nail Psoriasis Severity Index
Time to reach NAPSI=0 in the target nail | Up to Week 24
  Defined as time until NAPSI=0
Proportion of affected nails at baseline becoming nail Physician Global Assessment (PGA) responder at Week 24 | Baseline - Week 24
  Defined as Nail PGA response rate
Change from Baseline in Nail Psoriasis Visual Analogue Scale (VAS) Discomfort at Week 24 | Baseline - Week 24
  Defined as change in VAS
Patient Acceptance of Study Therapy at Week 24 | Baseline - Week 24
  Note: Missing values will be replaced with the worst score
Change from Baseline in EuroQoL-5Dimensions-5Levels (EQ-5D-5L) at Week 24 | Baseline - Week 24
  Defined as change in EQ-5D-5L
Change from Baseline in Dermatology Life Quality Index (DLQI) at Week 24 | Baseline - Week 24
  Defined as change in DLQI
Change from Baseline in Short Form 36 Health Survey (SF-36) at Week 24 | Baseline - Week 24
  Defined as change in SF-36
Change from Baseline in Nail Psoriasis Quality of Life Index (NPQ10) at Week 24 | Baseline - Week 24
  Defined as change in NPQ10

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Caserini, MD, Study Director — Polichem SA
Locations (58):
- United States (58):
  - Polichem Investigation Site no 47, Birmingham, Alabama
  - Polichem Investigation Site no 21, Phoenix, Arizona
  - Polichem Investigation Site no 11, Little Rock, Arkansas
  - Polichem Investigation Site no 45, North Hollywood, California
  - Polichem Investigation Site no 39, San Diego, California
  - Polichem Investigation Site no 56, Santa Monica, California
  - Polichem Investigation Site no 18, Washington D.C., District of Columbia
  - Polichem Investigation Site no 36, Clearwater, Florida
  - Polichem Investigation Site no 10, Miami, Florida
  - Polichem Investigation Site no 38, Miami, Florida
  - Polichem Investigation Site no 13, Miami, Florida
  - Polichem Investigation Site no 20, Miami Lakes, Florida
  - Polichem Investigation Site no 17, Ocala, Florida
  - Polichem Investigation Site no 35, Ormond Beach, Florida
  - Polichem Investigation site no 1, Tampa, Florida
  - Polichem Investigation Site no 24, Tampa, Florida
  - Polichem Investigation Site no 28, Tampa, Florida
  - Polichem Investigation Site no 25, Columbus, Georgia
  - Polichem Investigation Site no 23, Skokie, Illinois
  - Polichem Investigation Site no 29, West Dundee, Illinois
  - Polichem Investigation Site no 16, New Albany, Indiana
  - Polichem Investigation site no 3, West Des Moines, Iowa
  - Polichem Investigation Site no 22, Overland Park, Kansas
  - Polichem Investigation Site no 52, Louisville, Kentucky
  - Polichem Investigation Site no 19, Louisville, Kentucky
  - Polichem Investigation Site no 49, New Orleans, Louisiana
  - Polichem Investigation Site no 32, New Orleans, Louisiana
  - Polichem Investigation Site no 34, Rockville, Maryland
  - Polichem Investigation Site no 31, Ann Arbor, Michigan
  - Polichem Investigation Site no 2, Bay City, Michigan
  - Polichem Investigation Site no 9, Fridley, Minnesota
  - Polichem Investigation Site no 6, Omaha, Nebraska
  - Polichem Investigation Site no 5, Las Vegas, Nevada
  - Polichem Investigation Site no 41, Portsmouth, New Hampshire
  - Polichem Investigation Site no 58, East Windsor, New Jersey
  - Polichem Investigation Site no 54, Buffalo, New York
  - Polichem Investigation Site no 37, New York, New York
  - Polichem Investigation Site no 4, Rochester, New York
  - Polichem Investigation Site no 48, Rochester, New York
  - Polichem Investigation Site no 46, High Point, North Carolina
  - Polichem Investigation Site no 27, Winston-Salem, North Carolina
  - Polichem Investigation Site no 44, Cincinnati, Ohio
  - Polichem Investigation Site no 40, Norman, Oklahoma
  - Polichem Investigation Site no 14, Portland, Oregon
  - Polichem Investigation Site no 51, Johnston, Rhode Island
  - Polichem Investigation Site no 8, Charleston, South Carolina
  - Polichem Investigation Site no 26, Rapid City, South Dakota
  - Polichem Investigation Site no 12, Goodlettsville, Tennessee
  - Polichem Investigation Site no 7, Knoxville, Tennessee
  - Polichem Investigation Site no 56, Arlington, Texas
  - Polichem Investigation Site no 43, Dallas, Texas
  - Polichem Investigation Site no 42, Pflugerville, Texas
  - Polichem Investigation Site no 33, San Antonio, Texas
  - Polichem Investigation Site no 53, San Antonio, Texas
  - Polichem Investigation Site no 55, San Antonio, Texas
  - Polichem Investigation Site no 50, Murray, Utah
  - Polichem Investigation Site no 15, Norfolk, Virginia
  - Polichem Investigation Site no 30, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided